CLINICAL TRIAL: NCT05954533
Title: Cross Sectional Study to Determine Whether HEAVEN CRITERIA is a Better Tool Than Modified LEMON Score for Predicting Difficult Intubation in In-hospital Emergency Airway Management
Brief Title: HEAVEN CRITERIA vs Modified LEMON Score for Predicting Difficult Intubation
Status: Recruiting | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Dr Jaismol James, Junior Resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 39/22/IEC/JMMC&RI
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication
Keywords: HEAVEN criteria; Modified LEMON; Difficult airway; Prediction tool

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Emergency tracheal intubation is a lifesaving procedure frequently performed on critically ill and injured patients in the emergency department (ED). Emergency intubations are more difficult than elective intubations in the operating room setting because of the sicker patient population with a limited physiologic reserve and less controlled setting in the ED. Indeed, the proportion of difficult intubation ranges from 10% to 27% in the ED setting , whereas the rate ranges from 1% to 9% of elective intubation in the anaesthesia setting. Because emerging evidence demonstrates that repeated intubation attempts are associated with an increased risk of adverse events, early recognition of difficulty intubation with a systematic use of rescue methods in ED patients is critical. The commonest airway prediction tool is the LEMON score. In the modified LEMON score "Mallampati" was excluded as it was not a pragmatic assessment in the ED.

Existing difficult airway prediction tools were derived in the elective surgery environment and may not be applicable to emergency airway management. LEMON criteria was designed for preoperative clinical setting.

Hence in this study we are observing if HEAVEN (H- Hypoxemia E - extremes of age A - anatomical abnormalities V - vomit/ blood / fluid E - Exsanguination/anaemia N - neck mobility issues) is a better tool for predicting difficult intubatio.

ELIGIBILITY:
Inclusion Criteria:

* 1. All patients who undergo an endotracheal intubation in the emergency medicine department and 2. who legally give consent for the study or relatives give consent

Exclusion Criteria:

* Patients not consenting for the study or · Patients in cardio respiratory arrest

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from all age groups requiring endotracheal intubation and who gives consent for the study would be included.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
First attempt intubation success rate | Two hours
  First attempt success would be defined as the placement of an endotracheal tube in the trachea with a single insertion of a laryngoscope blade into the mouth and either a single insertion of an endotracheal tube into the mouth or a single insertion of a bougie into the mouth followed by a single insertion of an endotracheal tube into the mouth
Physicians assessment of intubation as easy or difficult | Two hours
  Physicians subjective assessment of airway as easy or difficult

SECONDARY OUTCOMES:
Total attempts of intubation. | Two hours
  Total number of attempts is divided into less than 10 number of attempts, 10 to 100 and >100attempts
Which criteria was the most frequent in causing difficult airway among HEAVEN | Two hours
Measuring if patient had hypotension | 2 hours
  SBP 100 and 20% decrease from baseline
Measuring if patient had hypertension | 2 hours
  SBP >160 and 20% increase from baseline
Measurement of bradycardia | Two hours
  Adults: HR < 40bpm and 20% decrease from baseline Paeds <12yrs: <60beats/min requiring atropine

CONTACTS AND LOCATIONS:
Overall Officials: DR APPU SUSEEL, MBBS,MD, Study Director — JMMCRI; DR SIJU V ABRAHAM, MBBS,MD, Study Director — JMMCRI
Locations (1):
- JMMCRI, Thrissur, Kerala, India